CLINICAL TRIAL: NCT00196027
Title: Feasibility Study of the PFX Closure System in Subjects With Cryptogenic Stroke, Transient Ischemia Attack or Paradoxical Embolism
Brief Title: Paradigm I Clinical Trial: Study of the PFX Closure System in Subjects With Cryptogenic Stroke, Transient Ischemia Attack or Paradoxical Embolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cierra (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-001 version 1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-11

CONDITIONS: Patent Foramen Ovale
MeSH Terms: conditions — Foramen Ovale, Patent

INTERVENTIONS:
Device: PFX Closure System

SUMMARY:
The primary objective of this study is to demonstrate the safety of the PFX Closure System when utilized for patients with patent foramen ovale (PFO) suffering from cryptogenic stroke, transient ischemic attacks or paradoxical embolism.

DETAILED DESCRIPTION:
Patent Foramen Ovale has been implicated in the etiology of paradoxical embolism, cryptogenic stroke, transient ischemic attack (TIA), and right to left gas embolism in severe decompression illness. An association between patent foramen ovale and severe migraine headaches has also been reported. Several implantable devices are being used for percutaneous closure of patent foramen ovale; we propose to use a non-implantable system to safely effect closure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 65 years old.
* Documented patent foramen ovale as determined by positive micro bubble study demonstrating right to left shunt and/or anatomic detection and functional assessment by pre-operative TCD and peri-operative echocardiography or ultrasound.
* Subjects with a history of cryptogenic stroke, transient ischemic attack or paradoxical embolism due to presumed paradoxical embolism through a PFO.
* Negative pregnancy test in women who are of child-bearing potential.
* Signed Informed Consent form.

Exclusion Criteria:

* Presence of thrombus at the intended site of closure, in left atrial appendage, or documented evidence of venous thrombus in the vessels through which access to the PFO is gained.
* Active endocarditis, or other infections producing a bacteremia.
* Presence of atrial septal defects or fenestrations which allow right-to-left shunting.
* Presence of implanted cardiac valves, pacemaker, implantable cardioverters/defibrillators (ICDs) or vena cava filters.
* Subjects with an intra-cardiac mass, tumor, clot or vegetation.
* Large, redundant atrial septal aneurysm that would prohibit adequate device access to the PFO or closure of the PFO, in the judgment of the investigator. A coexisting redundant atrial septal aneurysm is considered large if it prohibits the ability of the operator to adequately achieve vacuum suction necessary to achieve PFO closure.
* Presence of arrhythmia requiring pharmacologic or electrical therapy intervention or 1st degree block.
* Current enrollment in any investigational trial(s) using devices implanted in the vascular system or enrolled in any experimental drug study(ies) within three months of study entry.
* History of stroke or TIA within the past 14 days.
* Source of stroke other than paradoxical embolization.
* Hemodynamic instability or shock.
* Hypercoagulable disorder.
* Subjects with coagulation disorders who are unable to take antiplatelet or anticoagulant therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-04

PRIMARY OUTCOMES:
PFO closure as measured by transesophageal echocardiography (TEE) or transcranial Doppler (TCD) acutely post procedure

SECONDARY OUTCOMES:
PFO closure as measured by TEE or TCD at 30 days post procedure
Neurological death and adverse event (AE) rates for all subjects through 30 day follow-up
New arrhythmia rate through 30 day follow-up. For any subjects with new arrhythmia, arrhythmia status will also be evaluated at a follow-up visit from 3 to 6 months post procedure
PFO closure rate at 3 to 6 months for any subject not demonstrating complete closure at the 30 day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, MD, Principal Investigator — Cardio Vasculares Centrum - Sankt Katharien
Locations (1):
- CardioVascular Center, Sankt katharinen, Frankfurt am Main, Germany